CLINICAL TRIAL: NCT04773704
Title: Diagnostic Validity of a New Strategy for the Rapid Detection of Microorganisms and Their Resistance to Antibiotics Responsible for Pneumonia in Pediatric Intensive Care Units Using Protected Distal Samples
Brief Title: RAPid SOlution for Diagnosis of Respiratory Infection in Pediatric Intensive Care Unit
Acronym: RAPSODI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP20132
Record Dates: First submitted 2021-02-24; First posted 2021-02-26 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-02

CONDITIONS: Severe Infections Pneumonia With Invasive Ventilation in PICU
Keywords: Pneumonia; Pediatrics; Multiplex PCR; Mechanical ventilation
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FILMARRAY® Pneumonia Plus Panel technique — FILMARRAY® Pneumonia Plus Panel technique (multiplex PCR) on a respiratory sample
  Other Names: multiplex PCR

SUMMARY:
In patients with infectious pneumonitis, the FILMARRAY® Pneumonia Plus Panel technique (multiplex PCR) on a respiratory sample makes it possible to identify the responsible pathogen and its resistance to antibiotics in less than an hour and therefore to quickly adapt the anti- infectious. FILMARRAY® Pneumonia Plus has been validated on two types of specimens from adult intubated patients, tracheal aspirations and bronchoalveolar lavage. It has not been validated on protected distal samples which are nevertheless used in current practice. This project will study the diagnostic validity of this technique performed on this type of sample. If the validity is demonstrated, this will allow this technique to be used on the protected distal sample which is a reliable sample and used in the context of respiratory infections, in particular acquired under ventilation in children (bronchoalveolar lavage is less easy and little used in practice in children).

DETAILED DESCRIPTION:
In patients with infectious pneumonitis, the FILMARRAY® Pneumonia Plus Panel technique (multiplex PCR) on a respiratory sample makes it possible to identify the responsible pathogen and its resistance to antibiotics in less than an hour and therefore to quickly adapt the anti- infectious. FILMARRAY® Pneumonia Plus has been validated on two types of specimens from adult intubated patients, tracheal aspirations and bronchoalveolar lavage. It has not been validated on protected distal samples which are nevertheless used in current practice. This project will study the diagnostic validity of this technique performed on this type of sample. If the validity is demonstrated, this will allow this technique to be used on the protected distal sample which is a reliable sample and used in the context of respiratory infections, in particular acquired under ventilation in children (bronchoalveolar lavage is less easy and little used in practice in children).

As a result, this will allow a faster etiological diagnosis and adapted antibiotic therapy, guaranteeing better efficacy and a fairer antibiotic prescription.

Currently no studies concerning the FILMARRAY® Pneumonia Plus Panel are ongoing or have been performed with the protected distal samples.

This study would be innovative and unique in looking at its feasibility and validity on a type of sample used in current practice.

In addition, the use of a PCR-based technique allows a rapid microbiological diagnosis of lower respiratory infections under invasive mechanical ventilation, compared to the reference technique requiring 48 to 72 hours to give a definitive result.

This much shorter period allows for an appropriate antibiotic therapy early in the treatment, and potentially a reduction in ventilation and hospitalization times.

In addition, it detects antibiotic resistance genes allowing rapid identification of multi-resistant bacteria (resistant Staphylococcus aureus meticillin, enterobacteria producing ESBLs or carbapenemases) and thus adapting antibiotic therapy.

Our study will assess its diagnostic validity for the identification of the microorganisms responsible for pneumonia in intensive care and their resistance to antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in pediatric intensive care
* Patients under mechanical ventilation (intubated or tracheostomized)
* Age <18 years old

Exclusion Criteria:

* Contraindications to protected distal sampling
* Refusal to participate by at least one parent or legal guardian(s)
* Patient not covered by health insurance

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients hospitalized in pediatric intensive care unit, under mechanical ventilation (intubated or tracheostomized) with suspicion of infectious pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
concordance between the results of the FILMARRAY® Pneumonia on a protected distal sample (new strategy) and those obtained by culture and antibiogram (classic diagnosis, reference method) | 1 week
  Percentage of diagnostic agreement between the FilmArray result carried out on protected distal samples and the result of the reference method and description of the microorganisms most frequently found in cases of discrepancies.

SECONDARY OUTCOMES:
To establish the percentage of invalid analyzes on this type of sample. | 24 months
  Number of invalid analyzes out of the total number of analyzes performed on protected sample with the FilmArray.
Rate of true positives (agreement of positive results between new strategy and reference method) | 24 months
Rate of true negatives (agreement of negative results between new strategy and reference method). | 24 months
To establish the diagnostic time saving in real life use. | 24 months
  Differential in final rendering time between the new strategy and the reference method.
Number of diagnoses adjusted on the number of diagnoses sought in children whose sample was taken after antibiotic therapy. | 24 months
  Number of diagnoses adjusted on the number of diagnoses sought in children whose sample was taken after antibiotic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Robert Debré Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Geslain G, Cointe A, Naudin J, Dauger S, Poey N, Pages J, Le Roux E, Bonacorsi S. Diagnostic Accuracy of Blind Bronchial Sample Testing by BioFire Pneumonia plus Panel in Pediatric Intensive Care Unit Patients and Its Impact in Early Adaptation of Antimicrobial Therapy: A Prospective Observational Study. Pediatr Infect Dis J. 2024 Aug 1;43(8):725-730. doi: 10.1097/INF.0000000000004349. Epub 2024 Apr 8. PMID 38621162